CLINICAL TRIAL: NCT00076375
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Two Concentrations of Nanocrystalline Silver Cream (NPI) Applied Twice Daily in Adults With Mild to Moderate Atopic Dermatitis
Brief Title: Preliminary Study of Safety and Efficacy of Nanocrystalline Silver Cream in Atopic Dermatitis (Eczema)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nucryst Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 32101-2-01
Record Dates: First submitted 2004-01-21; First posted 2004-01-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-04

CONDITIONS: Atopic Dermatitis; Eczema
Keywords: Atopic Dermatitis; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

INTERVENTIONS:
Drug: Nanocrystalline silver cream (NPI)

SUMMARY:
Nanocrystalline silver (very small particles of silver) is the active ingredient in Acticoat dressings, which have been approved for the treatment of burns and other wounds. Silver has been used for decades as an effective antimicrobial agent. In animal studies, nanocrystalline silver cream (NPI) has also demonstrated anti-inflammatory activity. Thus, nanocrystalline silver cream is being evaluated in the treatment of inflammatory skin conditions such as atopic dermatitis (eczema).

Approximately 180 study subjects with a definitive diagnosis of mild to moderate eczema will be enrolled in this study. Subjects will be randomly assigned to treatment with placebo, 0.5% NPI or 1% NPI for the 6-week treatment period. Assessments of treatment effect and safety will be performed weekly. Upon completion of the study, subjects may be eligible for 12 weeks of open-label treatment with 1% NPI.

ELIGIBILITY:
* Male or female, any race, 18 to 65 years of age.
* Females must be post-menopausal, surgically sterile, or if of child-bearing potential, not pregnant (confirmed by test) and using an adequate method of birth control.
* Subjects must have eczema that covers a minimum of 5% total body surface area.
* Subjects must agree not to use other eczema medications for the 6-week study treatment period.
* Subjects must not be enrolled in another investigational drug study.
* Subjects must not be allergic to silver or cocoa butter.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-11; Study Completion 2004-04

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Radiant Research, Birmingham, Alabama
  - Medical Affliated Research Centers, Inc., Huntsville, Alabama
  - National Jewish Medical & Research Center, Denver, Colorado
  - nTouch Research, Washington D.C., District of Columbia
  - Radiant Research, West Palm Beach, Florida
  - Radiant Research, Boise, Idaho
  - Radiant Research, Overland Park, Kansas
  - Radiant Research, St Louis, Missouri
  - Sadick Dermatology & Aesthetic Surgery, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Clinical Research of Winston-Salem, Inc., Winston-Salem, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Radiant Research, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Radiant Research, Philadelphia, Pennsylvania
  - National Allergy, Asthma & Urticaria Centers of Charleston, P.A., Charleston, South Carolina
  - Radiant Research, Greer, South Carolina
  - ACE Research Specialists, Inc., Nashville, Tennessee
  - Radiant Research, Lakewood, Washington

REFERENCES:
- See also: Study sponsor's web site providing information about nanocrystalline silver. — http://www.nucryst.com
- See also: American Academy of Dermatology web site providing reference information on atopic dermatitis and other skin conditions. — http://www.aad.org
- See also: National Eczema Association web site providing resources and support to those with eczema. — http://www.nationaleczema.org